CLINICAL TRIAL: NCT04734639
Title: Appetite Response to Exercise- Versus Mixed (Exercise + Dietary Restriction)-Induced Energy Deficit in Adolescents With Obesity
Acronym: IDEX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Tza Nou - Maison médicale pour enfants et adolescentes (Unknown); Laboratoire AME2P (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2020 JULIAN 2; 2020-A03568-31 (Other: 2020-A03568-31)
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Obesity
Keywords: appetite control; obesity; Adolescents; exercise; Energy Deficit
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese adolescents (Experimental): 20 adolescents with obesity are involved and will perform the three conditions.
  Interventions: Behavioral: CON . control condition without exercise / rest condition; Behavioral: Def-Mixed. Condition with a mixed energy deficit induced by exercise + dietary restriction.; Behavioral: Def-EI. Condition with an energy-restriction energy deficit

INTERVENTIONS:
Behavioral: CON . control condition without exercise / rest condition — Control condition without exercise / rest condition. The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at dinner time. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
Behavioral: Def-Mixed. Condition with a mixed energy deficit induced by exercise + dietary restriction. — Def-Mixed. Condition with an exercise-induced energy deficit The adolescents will received a calibrated lundh meal with a deduction of 250 kcal compared with the lunch meal of Con; and will be asked to realise an acute exercise set at 65% of their capacities (cycling) during the afternoon, inducing an energy expenditure of 250 kcal. Dinner will be served ad libitum. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
Behavioral: Def-EI. Condition with an energy-restriction energy deficit — Condition with an energy-restriction energy deficit The adolescents will receive a calibrated breakfast reduced from 500 kcal compare to their CON and Def-mixed conditions. Dinner will be served ad libitum. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.

SUMMARY:
The aim of the present study is to compare the effect of iso-energetic energy deficits induced by energy restriction alone or exercise + dietary restriction (Mixed deficit) on energy intake and appetite feelings in adolescents with obesity.

DETAILED DESCRIPTION:
The present study will compare the nutritional response to an energy deficit of 500 kcal induced once by dietary restriction alone and once by a mixed deficit (50% by exercise and 50% by dietary restriction) (compared with a control condition). 18 adolescents with obesity will be asked to randomly complete three experimental sessions: i) one control session (CON); ii) one session with a dietary-induced energy deficit (Def-EI); iii) one session with a mixed deficit (50% by exercise and 50% by dietary restriction) (Def-Mixed).

Their ad libitum energy intake will be assessed at dinner time. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from different intervention of energy intake measured during an ad libitum buffet meal (in kcal). | day 1, day 8, day 15
  food intake will be measured ad libitum during a dinner buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Hunger feelings | day 1, day 8, day 15
  hunger area under the curve will be assessed using visual analogue scale through a the day
Food reward | day 1, day 8, day 15
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ) (Finlayson, King et al. 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Valérie JULIAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France